CLINICAL TRIAL: NCT04331964
Title: Dental Pulp Response to The Combination Use of Platelet-Rich Fibrin and Mineral Trioxide Aggregate in Partial Pulpotomy of Sound Human Premolars: A Randomized Controlled Trial
Brief Title: The Use of Platelet-Rich Fibrin in Partial Pulpotomy Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-OperDent-01-2020
Record Dates: First submitted 2020-03-29; First posted 2020-04-02 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Pulpitis
Keywords: Partial pulpotomy, platelet rich fibrin
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral Trioxide Aggregate (MTA) (Active Comparator): A standardized partial pulpotomy procedure will be performed after administration of local anesthesia. The exposed pulp tissues will be directly capped with a 3mm of MTA (Pro Root MTA) layer.
  Interventions: Procedure: partial pulpotomy
- MTA with platelet rich fibrin (PRF). (Experimental): A standardized partial pulpotomy procedure will be performed after administration of local anesthesia. The PRF membrane obtained after centrifugation of the patient's own blood is going to be placed over the exposed pulp. Then, a 3mm of MTA (Pro Root MTA) will be placed over the PRF membrane.
  Interventions: Procedure: partial pulpotomy

INTERVENTIONS:
Procedure: partial pulpotomy — Removal of a small portion of coronal pulp tissue after exposure, followed by application of a biomaterial directly onto the remaining pulp tissue prior to placement of a permanent restoration.

SUMMARY:
The aim of this study is to evaluate the clinical and histological pulp responses when MTA and a combined of MTA/PRF is used as pulp-capping agents after partial pulpotomy.

DETAILED DESCRIPTION:
Partial pulpotomy is generally considered as the treatment of choice for immature permanent teeth with reversible injury. Mineral trioxide aggregate (MTA) is a gold standard material as pulp capping agent in term of vital pulp therapy. Despite many advantages, MTA has a long setting time, little biological inductivity, difficult handling characteristics and high cost.

An essential aspect of tooth tissue engineering is the identification of a suitable scaffold to support cell growth and tissue regeneration. Platelet-Rich Fibrin (PRF) is a second generation platelet concentrate. It is strictly autologous and helps to release the growth factors necessary for the regeneration of dentin pulp complex. Therefore, PRF seems to be a suitable scaffold in vital pulp therapy.

Study sample, 24 intact maxillary or mandibular premolars which will be extracted for orthodontic reasons in 12 healthy volunteers. The sample will be chosen from the patients who are coming to the Orthodontic department in the Faculty of dentistry - Damascus university.

This study will be performed as split mouth study. For each selected patient, one premolar will be randomly allocated to MTA only and the other to combined MTA/PRF by a toss of coin. The main operator will give each patient a numerical code (from 1 to 12) whilst the teeth will have an alphabetical coding (e.g. For the patient coded as 1, premolar with MTA will be coded as 1-a, the other premolar with MTA/PRF will be coded as 1-b). In all patient documents, the teeth will be labeled in the same way so that the clinical examiner and a pathologist will be blinded to the capping technique used for each tooth whilst the main operator who perform a pulpotomy will know which technique is used for each premolar.

Postoperative pain and sensitivity to thermal stimuli will be analyzed after the treatment between two sides.

After 8 weeks, the teeth will be extracted and histologically evaluated in terms of inflammation, dentin bridge formation and its appearance.

ELIGIBILITY:
Inclusion Criteria:

1. No systemic disease and no medication consumption.
2. Participants, with healthy first premolars in either of the jaws, assigned for orthodontic extraction (scheduled extraction of the maxillary/mandibular premolars).
3. The premolar teeth needed to be fully erupted.
4. The premolar teeth needed to respond within the normal range to cold testing and heat testing.
5. The patients' parents had read, signed and thoroughly understood the informed consent.

Exclusion Criteria:

1. Presence of systematic disease and medication consumption of any type.
2. Anti-inflammatory medicine taken before and during the time of study.
3. Premolars with caries, restoration or any abnormality on periapical radiographs.
4. If the premolar teeth were not fully erupted.
5. If the premolar teeth revealed a lingering pain (a pain sensation that had the tendency to linger as a dull ache after the stimulus had been removed upon cold testing and heat testing).

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Thickness of dentin bridge | eight weeks after intervention
  This outcome will be evaluated by means of light microscopy linked to the camera with magnification of 4X, 20X, 40X and 100X. A periodontal probe will be placed over a histologic section to serve as a scale before image acquisition. The thickness of dentin bridge will be measured at the thickest, thinnest, and midmost point areas of the bridge. The average of the 3 values will be calculated. Each histologic section will be scored from 1-4, with 1 representing the most desired result and 4 representing the least desired result as follows:
  1. Thickness of dentin bridge is more than 0.25mm
  2. Thickness of dentin bridge is less than 0.25mm but more than 0.1mm.
  3. Thickness of dentin bridge is less than 0.1mm
  4. Partial or absent bridge.
Appearance of dentin bridge | eight weeks after intervention
  This outcome will be evaluated by means of light microscopy linked to the camera with magnification of 4X, 20X, 40X and 100X. Each histologic section will be scored from 1-4, with 1 representing the most desired result and 4 representing the least desired result as follows:
  1. Dentin that displays a tubular structure or dentin associated with irregular hard tissue that is not exhibit the characteristic tubular structure, but resemble bony tissue and often display cellular inclusions.
  2. Only irregular hard tissue deposition.
  3. Only a thin layer of hard tissue deposition.
  4. No hard tissue deposition
Intensity of Pulp Inflammation | eight weeks after intervention
  This outcome will be evaluated by means of light microscopy linked to the camera with magnification of 4X, 20X, 40X and 100X. Each histologic section will be scored from 1-4, with 1 representing the most desired result and 4 representing the least desired result as follows:
  1. Absent or very few inflammatory cells
  2. Mild: defined as an average of inflammatory cells is less than 10 cells.
  3. Moderate: defined as an average of inflammatory cells is more than10 cells but less than 25 cells.
  4. Severe: defined as an average of inflammatory cells is more than 25 cells.
Extension of Pulp Inflammation | eight weeks after intervention
  This outcome will be evaluated by means of light microscopy linked to the camera with magnification of 4X, 20X, 40X and 100X. Each histologic section will be scored from 1-4, with 1 representing the most desired result and 4 representing the least desired result as follows:
  1. Absent
  2. Mild: defined as inflammatory cells only next to pulp exposure site
  3. Moderate: defined as inflammatory cells observed in part of coronal pulp (in one-third or more of the coronal pulp or in the middle pulp)
  4. Severe: defined as all coronal pulp is infiltrated

SECONDARY OUTCOMES:
Postoperative pain: VAS | using a 0 to 10-cm visual analog scale (VAS) scale, pain will be record every 24 hours until the seventh day after intervention
  Patients or their parents will be asked to rate their pain by placing a mark on the line corresponding to their current level of postoperative pain. Pain on the VAS will be further categorized as no pain (0), or mild (1-3), moderate (4-6), or severe (7-10) pain.
Sensitivity to thermal stimuli | this outcome will be examined every week until the eighth week after intervention
  Cold testing will be performed with a refrigerant spray that apply to the tooth on a large cotton pellet. The responses will be further categorized as:
  * Normal response: patient's report that a sensation is felt but disappears immediately upon removal of the thermal stimulus.
  * Abnormal response: lingering or intensification of a painful sensation after the stimulus is removed, or an immediate, excruciatingly painful sensation as soon as the stimulus is placed on the tooth.
  * Lack of response to the stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Rami Zenaldeen, DDS MSc, Study Director — PhD student at the Endodontic and Operative Dentistry Department, University of Damascus Dental School, Damascus, Syrian Arab Republic; Ossama Aljabban, DDS MSc PhD, Principal Investigator — Professor at Endodontic and Operative Dentistry Department, University of Damascus Dental School, Damascus, Syrian Arab Republic; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor at Department of Orthodontics, University of Damascus Dental School, Damascus, Syrian Arab Republic
Locations (1):
- Department of Endodontics and Operative Dentistry, University of Damascus Dental School, Damascus, Syria, Damascus, Syria

REFERENCES:
- [Background] Azimi S, Fazlyab M, Sadri D, Saghiri MA, Khosravanifard B, Asgary S. Comparison of pulp response to mineral trioxide aggregate and a bioceramic paste in partial pulpotomy of sound human premolars: a randomized controlled trial. Int Endod J. 2014 Sep;47(9):873-81. doi: 10.1111/iej.12231. Epub 2014 Jan 13. PMID 24330490
- [Background] Bakhtiar H, Nekoofar MH, Aminishakib P, Abedi F, Naghi Moosavi F, Esnaashari E, Azizi A, Esmailian S, Ellini MR, Mesgarzadeh V, Sezavar M, About I. Human Pulp Responses to Partial Pulpotomy Treatment with TheraCal as Compared with Biodentine and ProRoot MTA: A Clinical Trial. J Endod. 2017 Nov;43(11):1786-1791. doi: 10.1016/j.joen.2017.06.025. Epub 2017 Aug 16. PMID 28822566
- [Background] Chailertvanitkul P, Paphangkorakit J, Sooksantisakoonchai N, Pumas N, Pairojamornyoot W, Leela-Apiradee N, Abbott PV. Randomized control trial comparing calcium hydroxide and mineral trioxide aggregate for partial pulpotomies in cariously exposed pulps of permanent molars. Int Endod J. 2014 Sep;47(9):835-42. doi: 10.1111/iej.12225. Epub 2014 Jan 28. PMID 24299006
- [Background] Hiremath H, Saikalyan S, Kulkarni SS, Hiremath V. Second-generation platelet concentrate (PRF) as a pulpotomy medicament in a permanent molar with pulpitis: a case report. Int Endod J. 2012 Jan;45(1):105-12. doi: 10.1111/j.1365-2591.2011.01973.x. Epub 2011 Nov 14. PMID 22077790
- [Background] Mehrvarzfar P, Abbott PV, Mashhadiabbas F, Vatanpour M, Tour Savadkouhi S. Clinical and histological responses of human dental pulp to MTA and combined MTA/treated dentin matrix in partial pulpotomy. Aust Endod J. 2018 Apr;44(1):46-53. doi: 10.1111/aej.12217. Epub 2017 Aug 18. PMID 28833942
- [Background] Solomon RV, Faizuddin U, Karunakar P, Deepthi Sarvani G, Sree Soumya S. Coronal Pulpotomy Technique Analysis as an Alternative to Pulpectomy for Preserving the Tooth Vitality, in the Context of Tissue Regeneration: A Correlated Clinical Study across 4 Adult Permanent Molars. Case Rep Dent. 2015;2015:916060. doi: 10.1155/2015/916060. Epub 2015 May 17. PMID 26097752
- [Background] Woo SM, Kim WJ, Lim HS, Choi NK, Kim SH, Kim SM, Jung JY. Combination of Mineral Trioxide Aggregate and Platelet-rich Fibrin Promotes the Odontoblastic Differentiation and Mineralization of Human Dental Pulp Cells via BMP/Smad Signaling Pathway. J Endod. 2016 Jan;42(1):82-8. doi: 10.1016/j.joen.2015.06.019. Epub 2015 Sep 9. PMID 26364004